CLINICAL TRIAL: NCT07091552
Title: Clinical Assessment of CAD/CAM Monolithic Complete Denture (Cross Over Controlled Clinical Trial)
Brief Title: Clinical Assessment of CAD/CAM Monolithic Complete Denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eman Assam (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Eman Assam, Assistant Lecturer of Prosthodontics, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 9208697
Record Dates: First submitted 2025-07-13; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Complete Denture

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM monolithic denture (Experimental)
  Interventions: Device: CAD/CAM monolithic denture
- Conventional denture (Active Comparator)
  Interventions: Device: Conventional denture

INTERVENTIONS:
Device: CAD/CAM monolithic denture — Based on the workflow suggested by the Ivoclar digital denture, conventional complete dentures will be scanned by using desktop scanner (Medit T710). The cameo and intaglio surfaces of the complete dentures will be scanned, and the scanned data will be exported as Standard Tessellation Language (STL) file to start the milling process.
  For the milling process, monolithic denture will be milled from a bicolored disk (Ivotion). One side is the denture base material made of high impact optimized polymethyl methacrylate (PMMA) while the other is the teeth material made of highly cross-linked PMMA with no filler. The bicolor disk is milled in a 5-axis milling machine in wet condition, through an uninterrupted milling process. Following the fast milling process the dentures will be finished and polished.
  Arms: CAD/CAM monolithic denture
Device: Conventional denture — The conventional set will be fabricated with the 5-appointment process: preliminary impressions (first appointment); definitive impressions (second appointment); interocclusal records and tooth selection (third appointment), the size of the teeth will be selected according to the library provided by 3Shape Dental System software to match the disc size; wax trial placement (fourth appointment); and denture adjustment and placement (fifth appointment). Conventional CD will be fabricated with the conventional lost wax technique and heat-polymerizing acrylic resin. The heat-polymerized CDs will be finished, and polished before placement. Adjustments will be made for the polished surface, tissue surface, borders, and occlusion. Occlusal errors will be adjusted through clinical remount of the finished dentures.
  Arms: Conventional denture

SUMMARY:
The aim of the study is to evaluate trueness, tooth position, retention, and patient satisfaction of CAD/CAM monolithic complete denture

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients, and willing to participate and sign the informed consent.
* No cognitive or psychological deficits.
* Moderate arch size with moderate undercut.
* No retrognathic or prognathic jaw relationship. (Normal horizontal ridge relationship)

Exclusion Criteria:

* Participants having undercuts, flabby ridge, severely resorbed ridges.
* Participants with noticeably poor neuromuscular control, hyposalivation, general health, or other issues rendering repeated appointments difficult.
* Oral mucosa exhibits papillary hyperplasia or pathologic changes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Trueness of CAD/CAM monolithic dentures | Baseline (Day 1)
  The CAD/CAM monolithic dentures will be scanned with laboratory scanner (Medit T710) . Data from the scans will be stored in a STL format. The scans of the conventional dentures will be considered the reference STL files. The scans of each denture base will be imported into an analytic software program. All the study denture file will be separated into cameo, and intaglio portions, according to the software program processing protocol. To determine the trueness (root mean square (RMS)), measured in mm of conventional and monolithic complete dentures, comparisons will be conducted for the cameo, and intaglio portions. All the study sample STL files will be superimposed to the corresponding reference STL files using voxel-based best-fit alignment in the surface matching software. Color maps will also be produced to demonstrate the qualitative three-dimensional differences between the test and reference files
Accuracy of tooth position | Baseline (Day 1)
  Accuracy will be verified by superimposing the tooth region data from the heat-cured and monolithic dentures on the tooth region data from the wax dentures using best fit algorithm of 3D data analytical software and measuring the displacement of the tooth arrangement. In addition, colour maps will be created using the 3D comparison function to visually display the direction and amount of tooth displacement. Using the software, a total of 48 measurement points will be established for maxillary dentures. Twenty-four measurement points will be defined on the anterior teeth: at the cusp tip or center of the incisal edge; at the mesio- and disto-incisal angles; and at the center of the lingual face of each tooth. Similarly, 24 measurement points will be defined on the posterior teeth at the cusp tips of each tooth. The average value of the dentures will be calculated for each of the 48 measurement points, and this will be used as the representative value of the measurement point.
Objective assessment of complete denture retention | Baseline (Day 1)
  Retention will be evaluated objectively by using digital force gauge that will be connected to a wire loop which is attached on the denture bases. This force will be measured in newtons (N) and recorded as the denture's retention. A total of 3 measurements will be made for each denture by the same investigator. The highest value will be recorded as the peak retention force and used for the analysis
Subjective assessment of complete denture retention | up to 6 months
  Complete dentures for each subject will be subjectively evaluated for denture retention by the use of the scoring system described by Kapur. Each denture is scored on a scale from 0 to 6 based on clinical examination:
  The total score (0-6) is used to classify denture performance as:
  Clinically poor: <6 Clinically fair: 6-8 Clinically good: >8
Patient satisfaction | up to 6 months
  A patient satisfaction questionnaire will be designed according to the Guckes questionnaires. Subjects will be asked eight questions that pertained to their satisfaction with their conventional or monolithic dentures. The responses: completely satisfied, partially satisfied, and dissatisfied were coded as 2, 1, and 0, respectively. The satisfaction variable was formed by adding the scores from the eight questions; the range was from 0 (very dissatisfied) to 16 (totally satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt